CLINICAL TRIAL: NCT02497911
Title: A Randomized Controlled Trial Comparing the Adductor Canal Catheter (ACC) and Intra-articular Catheter (IAC) Following Primary Total Knee Arthroplasty
Brief Title: A Trial Comparing Adductor Canal Catheter and Intraarticular Catheter Following Primary Total Knee Arthroplasty
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Principal Investigator, Jaime Baratta, Clinical Instructor, Thomas Jefferson University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 00002109
Record Dates: First submitted 2015-04-29; First posted 2015-07-15 (Estimated); Last update posted 2015-10-23 (Estimated); Status verified 2015-10

CONDITIONS: Acute Pain; Regional Anesthesia Morbidity
Keywords: Adductor Canal Catheter; Intraarticular Catheter; Arthroplasty, Replacement, Knee
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Adductor Canal Catheter (Experimental): Postoperatively, patients will be brought to the PACU. The needle insertion site, approximately 10cm proximal to their operative knee, will be exposed. A sterile field will be utilized and the femoral artery is identified with a high frequency linear transducer proximal to the operative knee. 18g insulated Tuohy needle will be inserted in an out-of-plane approach through the sartorius muscle to a final location in close proximity to the saphenous nerve. Once satisfied with needle placement and following negative aspiration, 15 cc's of 0.5% ropivicaine will be injected through the needle under visualization. A 20-g multi-orifice catheter will be inserted approximately 4 cm beyond the needle tip and secured.
  Interventions: Procedure: Adductor Canal Catheter; Drug: Ropivicaine
- Intraarticular Catheter (Experimental): Intra-articular catheters will be placed by the surgeon at the end of the procedure, before wound closure. A bupivacaine 0.5% infusion will be admin through the On-Q system and continued for 48 hours postoperatively.
  Interventions: Procedure: Intraarticular Catheter; Drug: Bupivicaine

INTERVENTIONS:
Procedure: Adductor Canal Catheter — 0.5% Ropivicaine for primary block and 0.2% Ropivicaine infusion by OnQ Pump
  Arms: Adductor Canal Catheter
Procedure: Intraarticular Catheter — 0.5% Bupivicaine for primary block and 0.125% Bupivicaine infusion by OnQ Pump
  Arms: Intraarticular Catheter
Drug: Ropivicaine
  Arms: Adductor Canal Catheter
Drug: Bupivicaine
  Arms: Intraarticular Catheter

SUMMARY:
The study is a prospective randomized controlled trial comparing intraarticular catheters and adductor canal catheters for postoperative analgesia following a primary Total Knee Arthroplasty (TKA).

DETAILED DESCRIPTION:
The study is a prospective, randomized controlled clinical trial comparing two methods of postoperative analgesia following primary TKA. Eligible primary TKA patients must be ASA I - III and require less than 20 mg oxycodone daily (or its equivalent). Exclusion criteria are: allergy to anesthetics, contraindication to regional anesthesia, sensory/motor disorder involving operative limb, non-english speaking, ASA IV or greater, psychiatric or cognitive disorders, incarceration, renal insufficiency with Cr > 2.0 and hepatic failure. When patients agree to participate in the study the following data will be collected by the research staff: ASA physical status, age, height, weight, gender, quantitative opiate use, numeric pain score with visual descriptors, painDETECT score (form included), WOMAC score (form included) and baseline Pain Management Questionnaire. When designated through randomization, intra-articular catheters will be placed intraoperatively by the surgeons, per usual protocol. ACC's will be placed postoperatively in the PACU. The catheters will exit the bandage in a similar fashion to blind the personnel collecting data, postoperatively. Those collecting data will not be blinded from identifying patients in the control group, as no catheter will exit the bandage. Potential risks for each procedure, which will be explained to the patient, include: bleeding, local infection, local anesthetic toxicity in the form of seizure and cardiac arrest and neuropathy. The preceding are commonly listed though infrequent complications of both procedures. Continuous ultrasound will guide the placement of the ACC.

ELIGIBILITY:
Inclusion Criteria:

* Age 40-85
* American Society of Anesthesiologists (ASA) Physical Status (PS) 1-3.
* Undergoing Unilateral, Primary, Total Knee Arthroplasty
* English as native language

Exclusion Criteria:

* Patient refusal
* History of opioid dependence
* Contraindication to peripheral nerve block
* Pre-existing significant neuropathy

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-11 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Post-operative pain | immediately postoperative period to post-operative day # 2
  postoperative pain as measured by Visual Analog Scale at rest and with movement

SECONDARY OUTCOMES:
Postoperative opioid consumption | immediat postoperative period to postoperative day # 2
  Opioid consumption within hospitalization
Chronic post-surgical pain | 6-8 weeks post-operative
  Assess post-surgical pain and function as measured by PainDetect and WOMAC questionnaires at 6-8 weeks post-operative compared to preoperative pain and function
Participation in Physical therapy | immediate postoperative period to postoperative day #2
  Physical therapy benchmarks such as active and passive range of motion

CONTACTS AND LOCATIONS:
Overall Officials: Jaime L Baratta, MD, Principal Investigator — Sidney Kimmel Medical Center at Thomas Jefferson University Hospital

REFERENCES:
- [Background] Fischer HB, Simanski CJ, Sharp C, Bonnet F, Camu F, Neugebauer EA, Rawal N, Joshi GP, Schug SA, Kehlet H; PROSPECT Working Group. A procedure-specific systematic review and consensus recommendations for postoperative analgesia following total knee arthroplasty. Anaesthesia. 2008 Oct;63(10):1105-23. doi: 10.1111/j.1365-2044.2008.05565.x. Epub 2008 Jul 10. PMID 18627367
- [Background] Charous MT, Madison SJ, Suresh PJ, Sandhu NS, Loland VJ, Mariano ER, Donohue MC, Dutton PH, Ferguson EJ, Ilfeld BM. Continuous femoral nerve blocks: varying local anesthetic delivery method (bolus versus basal) to minimize quadriceps motor block while maintaining sensory block. Anesthesiology. 2011 Oct;115(4):774-81. doi: 10.1097/ALN.0b013e3182124dc6. PMID 21394001
- [Background] Jenstrup MT, Jaeger P, Lund J, Fomsgaard JS, Bache S, Mathiesen O, Larsen TK, Dahl JB. Effects of adductor-canal-blockade on pain and ambulation after total knee arthroplasty: a randomized study. Acta Anaesthesiol Scand. 2012 Mar;56(3):357-64. doi: 10.1111/j.1399-6576.2011.02621.x. Epub 2012 Jan 4. PMID 22221014
- [Background] Kazak Bengisun Z, Aysu Salviz E, Darcin K, Suer H, Ates Y. Intraarticular levobupivacaine or bupivacaine administration decreases pain scores and provides a better recovery after total knee arthroplasty. J Anesth. 2010 Oct;24(5):694-9. doi: 10.1007/s00540-010-0970-x. Epub 2010 Jun 23. PMID 20571832
- [Background] Essving P, Axelsson K, Aberg E, Spannar H, Gupta A, Lundin A. Local infiltration analgesia versus intrathecal morphine for postoperative pain management after total knee arthroplasty: a randomized controlled trial. Anesth Analg. 2011 Oct;113(4):926-33. doi: 10.1213/ANE.0b013e3182288deb. Epub 2011 Aug 4. PMID 21821506